CLINICAL TRIAL: NCT06022185
Title: The Effect of Web-Based Education Given to Young Elders on E-Health Literacy, Digital Literacy and Healthy Lifestyle Levels
Brief Title: E-Health Literacy, Digital Literacy, Healthy Lifestyle and Web Based Education for Young Old Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Principal Investigator, Zeynep YILDIRIM, Teaching Assistant, Igdir University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Zeynep1
Record Dates: First submitted 2023-08-14; First posted 2023-09-01 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Healthy Lifestyle
Keywords: Elderly E-Health Digital Literacy Healthy Lifestyle

STUDY DESIGN:
Intervention Model Description: A total of 70 people, 35 in the experimental group and 35 in the control group, will be included in the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Web Based E-Health Literacy, Digital Literacy and Healthy Lifestyle Behaviors Training
  Interventions: Diagnostic Test: Web Based Training on E-health Literacy, Digital Literacy and Healthy Lifestyle Behaviors.
- Control Group (No Intervention): No action will be taken.

INTERVENTIONS:
Diagnostic Test: Web Based Training on E-health Literacy, Digital Literacy and Healthy Lifestyle Behaviors. — In the trainings planned for elderly individuals, digital literacy and e-health literacy levels will be improved, knowledge and awareness levels of elderly individuals will be increased and they will be provided with information in this direction. healthy lifestyle behaviors.
  Personal information form, "E-Health Literacy Scale", "Acquisition and Confirmation of Health Information in Digital Environment Scale", "Healthy Lifestyle Behaviors Scale-II" will be used in the research.
  Arms: Experimental group

SUMMARY:
A healthy lifestyle is defined as knowing and controlling all the behaviors that may affect the health of the individual and regulating his daily activities by choosing the appropriate behaviors for his/her own health status.

While many factors are effective on healthy lifestyle behaviors, health literacy is one of these factors. One of the health literacy measurement tools is e-health literacy.

E-health literacy is "the ability to search for, find, understand, evaluate health information from electronic sources and apply this information to addressing or solving a health problem.

Digital literacy is the ability of an individual to access, select, use, criticize and evaluate information in new and developing digital technologies. In this respect, the importance of digital literacy is an undeniable fact in the health sector and is thought to be related to e-health literacy.

In this direction, this research was planned to evaluate the effect of web-based education to be given to young and old individuals on e-health literacy, digital literacy and healthy lifestyle behaviors.

DETAILED DESCRIPTION:
A healthy lifestyle is defined as knowing and controlling all the behaviors that may affect the health of the individual and regulating his daily activities by choosing the appropriate behaviors for his/her own health status.

While many factors are effective on healthy lifestyle behaviors, health literacy is one of these factors. One of the health literacy measurement tools is e-health literacy.

E-health literacy is "the ability to search for, find, understand, evaluate health information from electronic sources and apply this information to addressing or solving a health problem.

Digital literacy is the ability of an individual to access, select, use, criticize and evaluate information in new and developing digital technologies. In this respect, the importance of digital literacy is an undeniable fact in the health sector and is thought to be related to e-health literacy.

In this direction, this research was planned to evaluate the effect of web-based education to be given to young and old individuals on e-health literacy, digital literacy and healthy lifestyle behaviors.

Material Method This study is a randomized controlled trial. The research is planned on young and old individuals registered to the family health center (FHC) in Iğdır city center between January 2023 and January 2025. The population of the research will consist of young and old individuals aged 65-74 who are registered in 2 FHCs selected by simple random sampling among 9 FHCs located in the city center of Iğdır. Based on previous similar studies to determine the sample size, it was calculated that there should be at least 31 individuals in each group as a result of the power analysis performed by taking the effect power =0.85, Alpha(α) =0.05, power 1- β (beta) =0.90. . However, considering the sample losses that may arise during the study, the number of samples was increased by 10% and a total of 70 people were planned, each group consisting of 35 people, by randomization.

Personal information form created by the researchers, "E-Health Literacy Scale", "Acquiring Health Information in Digital Environment and Confirmation Scale", "Healthy Lifestyle Behaviors Scale-II" will be used in the collection of research data.

Data Collection: The data will be encountered face-to-face by the researcher. Evaluation of Data: Data will be analyzed with SPSS for Windows 23 package program. In the analysis of the data, it is planned to use numbers, percentages, minimum and maximum values, mean and standard deviations, as well as the appropriate analysis techniques in the table below.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to Participate in Research
* Being between the ages of 65-74
* Being literate in Turkish
* Having a computer or mobile phone and internet connection at home
* Being able to use Whatsapp
* Not having a visual or auditory health problem that would prevent participation in the study.
* No communication barrier

Exclusion Criteria:

* Having a visual and auditory health problem that will prevent participation in the study.

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Pre-Test Data Collection | Time frame: One or two months
  The research pre-test data will be collected by the researcher between September 2023 and October 2023 by obtaining the contact information of the individuals registered and included in the study at Iğdır 14 Kasım Family Health Center and No. 1 Family Health Center.
  Persons in the experimental and control groups in the collection of data; "Personal Information Form", "E-Health Literacy Scale", "Acquiring Health Information in Digital Environment and Confirmation Scale", "Healthy Lifestyle Behaviors Scale-II" will be applied. For the e-Health Literacy Scale The highest score is 40 and the lowest score is 8. The highest score that can be obtained for the Healthy Lifestyle Behaviors Scale II (SYBDS II) is 52, and the lowest score is 208.
  The score obtained from the Scale for Obtaining and Confirming Health Information in the Digital Environment is between 1 and 5 is changing
Collection of Post-Test Data | Time frame: one or two months
  For the experimental group, training videos related to the topics prepared in line with the training guide will be prepared every week for 6 weeks and uploaded to the web system and shared on whatsapp at the same time. Feedback will be received by creating interactive communication environments.After the trainings are over, the post-test data will be collected after a total of 1 and a half months without any follow-up process.
  It is planned to collect the post-test data between November 2023 and December 2023 in Iğdır 14 Kasım Family Health Center.Persons in the experimental and control groups in the collection of data; "Personal Information Form", "E-Health Literacy Scale", "Acquiring Health Information in Digital Environment and Confirmation Scale", "Healthy Lifestyle Behaviors Scale-II" will be applied.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep YILDIRIM, Doctorate, Principal Investigator — Igdir University
Locations (1):
- Igdir University, Iğdır, Turkey (Türkiye)